CLINICAL TRIAL: NCT01218126
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-centre, Dose Ranging Study to Evaluate the Efficacy and Safety of Losmapimod (GW856553) Tablets Administered Twice Daily Compared With Placebo for 24 Weeks in Adult Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-centre, Dose Ranging Study to Evaluate the Efficacy and Safety of Losmapimod Tablets Administered Twice Daily Compared With Placebo for 24 Weeks in Adult Subjects With Chronic Obstructive Pulmonary Disease (COPD).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113006
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- losmapimod 2.5 mg (Experimental): losmapimod 2.5 mg
  Interventions: Drug: losmapimod
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- losmapimod 7.5 mg (Experimental): losmapimod 7.5 mg
  Interventions: Drug: losmapimod
- losmapimod 15 mg (Experimental): losmapimod 15 mg
  Interventions: Drug: losmapimod

INTERVENTIONS:
Drug: losmapimod — comparison of different dosages of drug 2.5 mg, 7.5 mg or 15 mg
  Arms: losmapimod 15 mg; losmapimod 2.5 mg; losmapimod 7.5 mg
Drug: placebo — placebo comparison with active
  Arms: placebo

SUMMARY:
Randomised, double-blind, parallel-group, multi-centre study evaluating three doses of losmapimod (2.5mg, 7.5 mg and 15 mg) twice daily (BID) versus placebo on exercise tolerance. Eligible subjects will be randomised to treatment after a one-week run-in period. The duration of the treatment period is 24 weeks. An estimated 1000 subjects will be screened to reach the target enrolment of approximately 600 randomised subjects.

ELIGIBILITY:
Inclusion Criteria:

* clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society
* FEV1/FVC ratio of ≤0.70
* FEV1 ≤ 80% of predicted normal
* 6MWD < 350m
* male or female outpatients aged ≥40 years of age
* current or prior history of ≥10 pack-years of cigarette smoking
* aspartate transaminase (AST) or alanine transaminase (ALT) <2x Upper Limit Normal (ULN)
* alkaline phosphatase (alk phos), and bilirubin <1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* QTc <450 msec* on baseline ECG. For subjects with baseline complete bundle branch block, the QTc must be <480msec* on baseline ECG.

Exclusion Criteria:

* current diagnosis of asthma
* pregnant or lactating
* α1-antitrypsin deficiency
* lung resection
* chest X-ray (or CT scan) that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD
* exacerbation of COPD within previous 12 weeks
* treatment with roflumilast within previous 2 weeks and throughout the treatment period
* lower respiratory tract infection that required the use of antibiotics within previous 12 weeks
* long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day
* participation in the acute phase of a Pulmonary Rehabilitation Program within 12 weeks or planned during the study
* carcinoma that has not been in complete remission for at least 5 years
* current or chronic history of liver disease
* positive Hepatitis B surface antigen or positive Hepatitis C antibody
* Body Mass Index (BMI) > 35
* known or suspected history of alcohol or drug abuse within the last 2 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2010-11-04 (Actual); Primary Completion 2011-12-21 (Actual); Study Completion 2011-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (37):
- United States (8):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Richmond, Virginia
- Argentina (5):
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Czechia (4):
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Zlín
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (8):
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Rüsselsheim am Main, Hesse
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Norway (6):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Follebu
  - GSK Investigational Site, Harstad
  - GSK Investigational Site, Levanger
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Trondheim
- GSK Investigational Site, Seoul, South Korea
- Ukraine (3):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Largajolli A, Beerahee M, Yang S. Bayesian approach to investigate a two-state mixed model of COPD exacerbations. J Pharmacokinet Pharmacodyn. 2019 Aug;46(4):371-384. doi: 10.1007/s10928-019-09643-6. Epub 2019 Jun 13. PMID 31197640
- [Derived] Watz H, Barnacle H, Hartley BF, Chan R. Efficacy and safety of the p38 MAPK inhibitor losmapimod for patients with chronic obstructive pulmonary disease: a randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2014 Jan;2(1):63-72. doi: 10.1016/S2213-2600(13)70200-5. Epub 2013 Dec 5. PMID 24461903
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 04 November 2010 to 22 December 2011 across 65 centers worldwide. A total of 1000 participants with history of COPD exacerbations were planned to be screened and finally, 600 participants were planned to be randomized.
Pre-assignment Details: A total of 886 participants were screened, 282 were screen failures, remaining 604 were randomized to receive the study drug. Out of the randomized 604, 2 participants did not receive the study drug due to error in randomization.
Groups:
- Placebo: Participants received placebo matching Losmapimod tablet twice daily orally for a period of 24 weeks. During the run-in and treatment periods all participants continued their existing COPD therapy at a constant dose, including long-acting β2-agonists (LABA); long-acting muscarinic antagonists (LAMA); xanthines and/or inhaled corticosteroids (ICS). Participants were followed-up for 1 week after the last dose of the study drug.
- Losmapimod 2.5 mg: Participants received Losmapimod 2.5 milligram (mg) tablet twice daily orally for a period of 24 weeks. During the run-in and treatment periods all participants continued their existing COPD therapy at a constant dose, including long-acting β2-agonists (LABA); long-acting muscarinic antagonists (LAMA); xanthines and/or inhaled corticosteroids (ICS). Participants were followed-up for 1 week after the last dose of the study drug.
- Losmapimod 7.5 mg: Participants received Losmapimod 7.5 mg tablet twice daily orally for a period of 24 weeks. During the run-in and treatment periods all participants continued their existing COPD therapy at a constant dose, including long-acting β2-agonists (LABA); long-acting muscarinic antagonists (LAMA); xanthines and/or inhaled corticosteroids (ICS). Participants were followed-up for 1 week after the last dose of the study drug.
- Losmapimod 15 mg: Participants received Losmapimod 7.5 mg tablet twice daily orally for 4 weeks followed by Losmapimod 15 mg for a total period of 24 weeks. During the run-in and treatment periods all participants continued their existing COPD therapy at a constant dose, including long-acting β2-agonists (LABA); long-acting muscarinic antagonists (LAMA); xanthines and/or inhaled corticosteroids (ICS). Participants were followed-up for 1 week after the last dose of the study drug.
Period: Overall Study
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
Started | 153 | 149 | 151 | 149
Completed | 129 | 127 | 127 | 114
Not Completed | 24 | 22 | 24 | 35
Not completed — Adverse Event | 8 | 10 | 12 | 16
Not completed — Lack of Efficacy | 7 | 2 | 2 | 6
Not completed — Protocol Violation | 5 | 2 | 2 | 3
Not completed — Protocol-defined stopping criteria | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Physician Decision | 1 | 2 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 5 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Losmapimod 2.5 mg: Participants received Losmapimod 2.5 mg tablet twice daily orally for a period of 24 weeks. During the run-in and treatment periods all participants continued their existing COPD therapy at a constant dose, including long-acting β2-agonists (LABA); long-acting muscarinic antagonists (LAMA); xanthines and/or inhaled corticosteroids (ICS). Participants were followed-up for 1 week after the last dose of the study drug.
- Total: Total of all reporting groups
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg | Total
Number analyzed (Participants) | 153 | 149 | 151 | 149 | 602
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (8.64) | 66.1 (8.64) | 66.1 (7.76) | 64.8 (9.26) | 65.2 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 48 | 44 | 189
  Male | 104 | 101 | 103 | 105 | 413
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 19 | 16 | 18 | 23 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 1 | 8 | 14
  White | 131 | 131 | 132 | 118 | 512
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Six Minute Walk Distance (6MWD) at Week 4, 12 and 24
Description: Exercise tolerance was assessed using the 6MWD. If a participant was recorded as having used supplemental oxygen or a walking aid (including sitting down then continuing walking) or a technical problem during a 6MWD then that walk was considered as invalid; otherwise the 6MWD was considered as valid. The baseline 6MWD value was defined as the longest distance walked, for a valid walk, at Visit 2. Variability between the distances walked during the first six-minute walk test (6MWD1) and the second six-minute walk test (6MWD2) being compared was defined as: Variability = [100 x (6MWD2 - 6MWD1)]/6MWD1. Change from Baseline was calculated as the endpoint value minus the Baseline value. Baseline visit was Visit 2 (Week 0).
Time Frame: Baseline (Week 0) and Week 4, 12, 24
Population: Intent-to-treat (ITT) population consisted of all participants randomized to treatment and who received at least one dose of study drug. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Meter (m)
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
Number analyzed (Participants) | 153 | 149 | 151 | 149
Meter (m)
  Week 4: number analyzed (Participants) | 145 | 140 | 145 | 141
  Week 4 | 314.4 (2.79) | 311.8 (2.84) | 313.2 (2.78) | 319.9 (2.83)
  Week 12: number analyzed (Participants) | 135 | 132 | 137 | 124
  Week 12 | 321.6 (3.53) | 322.2 (3.58) | 320.2 (3.50) | 323.4 (3.65)
  Week 24: number analyzed (Participants) | 129 | 126 | 132 | 120
  Week 24 | 330.6 (4.13) | 324.0 (4.19) | 325.9 (4.09) | 327.2 (4.27)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 4; Test type: Superiority or Other; p = 0.517, mixed model repeated measures; Mean Difference (Net) = -2.6, 95% CI 2-sided [-10.4 to 5.2] — Analysis performed using a repeated measures model with covariates of treatment, region, smoking status at screening (stratum), history of exacerbations, baseline, visit, visit by baseline and visit by treatment interactions
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 4; Test type: Superiority or Other; p = 0.763, mixed model repeated measures; Mean Difference (Net) = -1.2, 95% CI 2-sided [-8.9 to 6.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 4; Test type: Superiority or Other; p = 0.164, mixed model repeated measures; Mean Difference (Net) = 5.5, 95% CI 2-sided [-2.3 to 13.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 12; Test type: Superiority or Other; p = 0.900, mixed model repeated measures; Mean Difference (Net) = 0.6, 95% CI 2-sided [-9.2 to 10.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 12; Test type: Superiority or Other; p = 0.788, mixed model repeated measures; Mean Difference (Net) = -1.3, 95% CI 2-sided [-11.1 to 8.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 12; Test type: Superiority or Other; p = 0.722, mixed model repeated measures; Mean Difference (Net) = 1.8, 95% CI 2-sided [-8.2 to 11.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 24; Test type: Superiority or Other; p = 0.260, mixed model repeated measures; Mean Difference (Net) = -6.7, 95% CI 2-sided [-18.2 to 4.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 24; Test type: Superiority or Other; p = 0.422, mixed model repeated measures; Mean Difference (Net) = -4.7, 95% CI 2-sided [-16.1 to 6.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 24; Test type: Superiority or Other; p = 0.564, mixed model repeated measures; Mean Difference (Net) = -3.4, 95% CI 2-sided [-15.1 to 8.2] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Sec (FEV1) at Week 4, 8, 12, 16, 20 and 24
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Pre and post-bronchodilator spirometry was performed by the investigator. For post-bronchodilator measurements, spirometry was performed 10-15 minutes after inhalation of 400/360 microgram (mcg) of salbutamol/albuterol. Participants were asked to withhold all bronchodilator therapy (regularly used ipratropium bromide and salbutamol/albuterol used as required) for at least 4 hours prior to spirometric testing. The change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization values.Baseline visit was Visit 2 (Week 0).
Time Frame: Baseline(Week 0) and Week 4, 8, 12, 16, 20 and 24
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millilitre(mL)
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
Number analyzed (Participants) | 153 | 149 | 151 | 149
Millilitre(mL)
  Pre-Bronchodilator Week 4: number analyzed (Participants) | 147 | 141 | 146 | 141
  Pre-Bronchodilator Week 4 | 2 (13.6) | 1 (13.9) | -5 (13.7) | 30 (13.9)
  Pre-Bronchodilator Week 8: number analyzed (Participants) | 143 | 138 | 145 | 131
  Pre-Bronchodilator Week 8 | 9 (15.2) | 7 (15.4) | 17 (15.1) | 45 (15.7)
  Pre-Bronchodilator Week 12: number analyzed (Participants) | 135 | 132 | 134 | 126
  Pre-Bronchodilator Week 12 | -15 (15.0) | 1 (15.2) | 4 (15.0) | 34 (15.5)
  Pre-Bronchodilator Week 16: number analyzed (Participants) | 133 | 132 | 137 | 126
  Pre-Bronchodilator Week 16 | -7 (15.4) | 15 (15.6) | 18 (15.3) | 17 (15.9)
  Pre-Bronchodilator Week 20: number analyzed (Participants) | 132 | 132 | 131 | 117
  Pre-Bronchodilator Week 20 | -13 (15.5) | -7 (15.6) | 20 (15.5) | 16 (16.2)
  Pre-Bronchodilator Week 24: number analyzed (Participants) | 128 | 127 | 127 | 117
  Pre-Bronchodilator Week 24 | -1 (15.2) | 3 (15.3) | 17 (15.2) | 14 (15.8)
  Post-Bronchodilator Week 4: number analyzed (Participants) | 147 | 141 | 146 | 140
  Post-Bronchodilator Week 4 | -2 (12.8) | 3 (13.1) | 14 (12.8) | 30 (13.1)
  Post-Bronchodilator Week 8: number analyzed (Participants) | 142 | 137 | 145 | 130
  Post-Bronchodilator Week 8 | 8 (15.7) | 7 (16.0) | 14 (15.6) | 51 (16.3)
  Post-Bronchodilator Week 12: number analyzed (Participants) | 135 | 132 | 133 | 125
  Post-Bronchodilator Week 12 | -1 (15.8) | -11 (16.0) | 9 (15.8) | 37 (6.3)
  Post-Bronchodilator Week 16: number analyzed (Participants) | 133 | 132 | 136 | 126
  Post-Bronchodilator Week 16 | 1 (15.4) | -6 (15.6) | 20 (15.3) | 27 (15.9)
  Post-Bronchodilator Week 20: number analyzed (Participants) | 132 | 132 | 131 | 117
  Post-Bronchodilator Week 20 | -4 (15.4) | -22 (15.6) | 23 (15.4) | 10 (16.1)
  Post-Bronchodilator Week 24: number analyzed (Participants) | 127 | 126 | 127 | 117
  Post-Bronchodilator Week 24 | 3 (15.6) | -6 (15.7) | 24 (15.6) | 10 (16.1)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 4; Test type: Superiority or Other; p = 0.968, mixed model repeated measures; Mean Difference (Net) = -1, 95% CI 2-sided [-39 to 38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FEV1 Placebo versus Losmapimod 7.5 mg at Week 4; Test type: Superiority or Other; p = 0.715, mixed model repeated measures; Mean Difference (Net) = -7, 95% CI 2-sided [-45 to 31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 4; Test type: Superiority or Other; p = 0.152, mixed model repeated measures; Mean Difference (Net) = 28, 95% CI 2-sided [-10 to 66] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 8; Test type: Superiority or Other; p = 0.922, mixed model repeated measures; Mean Difference (Net) = -2, 95% CI 2-sided [-45 to 40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 8; Test type: Superiority or Other; p = 0.694, mixed model repeated measures; Mean Difference (Net) = 8, 95% CI 2-sided [-34 to 50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 8; Test type: Superiority or Other; p = 0.094, mixed model repeated measures; Mean Difference (Net) = 37, 95% CI 2-sided [-6.3 to 79] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 12; Test type: Superiority or Other; p = 0.456, mixed model repeated measures; Mean Difference (Net) = 16, 95% CI 2-sided [-26 to 58] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 12; Test type: Superiority or Other; p = 0.355, mixed model repeated measures; Mean Difference (Net) = 20, 95% CI 2-sided [-22 to 61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 12; Test type: Superiority or Other; p = 0.023, mixed model repeated measures; Mean Difference (Net) = 49, 95% CI 2-sided [6.7 to 91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 16; Test type: Superiority or Other; p = 0.320, mixed model repeated measures; Mean Difference (Net) = 22, 95% CI 2-sided [-21 to 65] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 16; Test type: Superiority or Other; p = 0.267, mixed model repeated measures; Mean Difference (Net) = 24, 95% CI 2-sided [-19 to 67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 16; Test type: Superiority or Other; p = 0.289, mixed model repeated measures; Mean Difference (Net) = 24, 95% CI 2-sided [-20 to 67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 20; Test type: Superiority or Other; p = 0.786, mixed model repeated measures; Mean Difference (Net) = 6, 95% CI 2-sided [-37 to 49] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 20; Test type: Superiority or Other; p = 0.134, mixed model repeated measures; Mean Difference (Net) = 33, 95% CI 2-sided [-10 to 76] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 20; Test type: Superiority or Other; p = 0.191, mixed model repeated measures; Mean Difference (Net) = 29, 95% CI 2-sided [-15 to 74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 24; Test type: Superiority or Other; p = 0.852, mixed model repeated measures; Mean Difference (Net) = 4, 95% CI 2-sided [-38 to 46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 24; Test type: Superiority or Other; p = 0.397, mixed model repeated measures; Mean Difference (Net) = 18, 95% CI 2-sided [-24 to 60] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 24; Test type: Superiority or Other; p = 0.494, mixed model repeated measures; Mean Difference (Net) = 15, 95% CI 2-sided [-28 to 58] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 4; Test type: Superiority or Other; p = 0.807, mixed model repeated measures; Mean Difference (Net) = 4, 95% CI 2-sided [-31 to 40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 4; Test type: Superiority or Other; p = 0.386, mixed model repeated measures; Mean Difference (Net) = 16, 95% CI 2-sided [-20 to 51] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 4; Test type: Superiority or Other; p = 0.089, mixed model repeated measures; Mean Difference (Net) = 31, 95% CI 2-sided [-4.8 to 67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 8; Test type: Superiority or Other; p = 0.958, mixed model repeated measures; Mean Difference (Net) = -1, 95% CI 2-sided [-45 to 43] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 8; Test type: Superiority or Other; p = 0.766, mixed model repeated measures; Mean Difference (Net) = 7, 95% CI 2-sided [-37 to 50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 8; Test type: Superiority or Other; p = 0.060, mixed model repeated measures; Mean Difference (Net) = 43, 95% CI [-1.7 to 87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 12; Test type: Superiority or Other; p = 0.678, mixed model repeated measures; Mean Difference (Net) = -9, 95% CI 2-sided [-53 to 35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 12; Test type: Superiority or Other; p = 0.636, mixed model repeated measures; Mean Difference (Net) = 11, 95% CI 2-sided [-33 to 54] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 12; Test type: Superiority or Other; p = 0.094, mixed model repeated measures; Mean Difference (Net) = 38, 95% CI 2-sided [-6.5 to 83] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 16; Test type: Superiority or Other; p = 0.772, mixed model repeated measures; Mean Difference (Net) = -6, 95% CI 2-sided [-49 to 37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 29: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 16; Test type: Superiority or Other; p = 0.387, mixed model repeated measures; Mean Difference (Net) = 19, 95% CI 2-sided [-24 to 61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 30: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 16; Test type: Superiority or Other; p = 0.243, mixed model repeated measures; Mean Difference (Net) = 26, 95% CI 2-sided [-18 to 69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 31: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 20; Test type: Superiority or Other; p = 0.398, mixed model repeated measures; Mean Difference (Net) = -19, 95% CI 2-sided [-62 to 25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 32: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 20; Test type: Superiority or Other; p = 0.214, mixed model repeated measures; Mean Difference (Net) = 27, 95% CI 2-sided [-16 to 70] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 33: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 20; Test type: Superiority or Other; p = 0.526, mixed model repeated measures; Mean Difference (Net) = 14, 95% CI 2-sided [-30 to 58] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 34: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 2.5 mg at Week 24; Test type: Superiority or Other; p = 0.671, mixed model repeated measures; Mean Difference (Net) = -9, 95% CI 2-sided [-53 to 34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 35: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 7.5 mg at Week 24; Test type: Superiority or Other; p = 0.355, mixed model repeated measures; Mean Difference (Net) = 20, 95% CI 2-sided [-23 to 64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 36: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FEV1 for Placebo versus Losmapimod 15 mg at Week 24; Test type: Superiority or Other; p = 0.781, mixed model repeated measures; Mean Difference (Net) = 6, 95% CI 2-sided [-38 to 50] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Week 4, 8, 12, 16, 20 and 24
Description: FVC is the total amount of air exhaled during the lung function test. and post-bronchodilator spirometry was performed by the investigator. For post-bronchodilator measurements, spirometry was performed 10-15 minutes after inhalation of 400/360 microgram (mcg) of salbutamol/albuterol. Participants were asked to withhold all bronchodilator therapy (regularly used ipratropium bromide and salbutamol/albuterol used as required) for at least 4 hours prior to spirometric testing. The change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization values.. Baseline visit was Visit 2 (Week 0).
Time Frame: Baseline(Week 0) and Week 4, 8, 12, 16, 20 and 24
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
Number analyzed (Participants) | 153 | 149 | 151 | 149
mL
  Pre-Bronchodilator Week 4: number analyzed (Participants) | 147 | 141 | 146 | 141
  Pre-Bronchodilator Week 4 | -24 (28.3) | -11 (28.9) | -55 (28.3) | 33 (28.9)
  Pre-Bronchodilator Week 8: number analyzed (Participants) | 143 | 138 | 145 | 131
  Pre-Bronchodilator Week 8 | 8 (29.8) | -2 (30.4) | -5 (29.6) | 54 (30.9)
  Pre-Bronchodilator Week 12: number analyzed (Participants) | 135 | 132 | 134 | 126
  Pre-Bronchodilator Week 12 | -50 (31.4) | -5 (31.8) | -34 (31.3) | 25 (32.4)
  Pre-Bronchodilator Week 16: number analyzed (Participants) | 133 | 132 | 137 | 126
  Pre-Bronchodilator Week 16 | -34 (32.3) | -24 (32.6) | -9 (32.0) | 8 (33.3)
  Pre-Bronchodilator Week 20: number analyzed (Participants) | 132 | 132 | 131 | 117
  Pre-Bronchodilator Week 20 | -20 (31.9) | -51 (32.2) | -13 (31.9) | 13 (33.4)
  Pre-Bronchodilator Week 24: number analyzed (Participants) | 128 | 127 | 127 | 117
  Pre-Bronchodilator Week 24 | -18 (32.1) | -41 (32.4) | -25 (32.1) | 25 (33.4)
  Post-Bronchodilator Week 4: number analyzed (Participants) | 147 | 141 | 146 | 140
  Post-Bronchodilator Week 4 | -36 (25.8) | -29 (26.3) | -24 (25.8) | 35 (26.4)
  Post-Bronchodilator Week 8: number analyzed (Participants) | 142 | 137 | 145 | 130
  Post-Bronchodilator Week 8 | 3 (29.2) | -22 (29.7) | -27 (29.0) | 69 (30.3)
  Post-Bronchodilator Week 12: number analyzed (Participants) | 135 | 132 | 133 | 125
  Post-Bronchodilator Week 12 | -23 (31.2) | -34 (31.6) | -10 (31.2) | 52 (32.2)
  Post-Bronchodilator Week 16: number analyzed (Participants) | 133 | 132 | 136 | 126
  Post-Bronchodilator Week 16 | -17 (31.0) | -48 (31.4) | -1 (30.8) | 55 (32.0)
  Post-Bronchodilator Week 20: number analyzed (Participants) | 132 | 132 | 131 | 117
  Post-Bronchodilator Week 20 | -14 (31.2) | -78 (31.5) | -26 (31.1) | 35 (32.6)
  Post-Bronchodilator Week 24: number analyzed (Participants) | 127 | 126 | 127 | 117
  Post-Bronchodilator Week 24 | -15 (31.2) | -43 (31.5) | -5 (31.2) | 20 (32.4)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 4; Test type: Superiority or Other; p = 0.742, mixed model repeated measures; Mean Difference (Net) = 13, 95% CI 2-sided [-66 to 93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 4; Test type: Superiority or Other; p = 0.446, mixed model repeated measures; Mean Difference (Net) = -30, 95% CI 2-sided [-109 to 48] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 4; Test type: Superiority or Other; p = 0.157, mixed model repeated measures; Mean Difference (Net) = 57, 95% CI 2-sided [-22 to 137] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 8; Test type: Superiority or Other; p = 0.826, mixed model repeated measures; Mean Difference (Net) = -9, 95% CI 2-sided [-93 to 74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 8; Test type: Superiority or Other; p = 0.773, mixed model repeated measures; Mean Difference (Net) = -12, 95% CI [-95 to 70] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 8; Test type: Superiority or Other; p = 0.277, mixed model repeated measures; Mean Difference (Net) = 47, 95% CI 2-sided [-38 to 131] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 12; Test type: Superiority or Other; p = 0.319, mixed model repeated measures; Mean Difference (Net) = 45, 95% CI 2-sided [-43 to 132] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 12; Test type: Superiority or Other; p = 0.716, mixed model repeated measures; Mean Difference (Net) = 16, 95% CI 2-sided [-71 to 103] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 12; Test type: Superiority or Other; p = 0.098, mixed model repeated measures; Mean Difference (Net) = 75, 95% CI 2-sided [-14 to 163] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 16; Test type: Superiority or Other; p = 0.832, mixed model repeated measures; Mean Difference (Net) = 10, 95% CI 2-sided [-80 to 100] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 16; Test type: Superiority or Other; p = 0.579, mixed model repeated measures; Mean Difference (Net) = 25, 95% CI 2-sided [-64 to 114] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 16; Test type: Superiority or Other; p = 0.369, mixed model repeated measures; Mean Difference (Net) = 42, 95% CI 2-sided [-49 to 133] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 20; Test type: Superiority or Other; p = 0.487, mixed model repeated measures; Mean Difference (Net) = -32, 95% CI 2-sided [-121 to 58] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 20; Test type: Superiority or Other; p = 0.887, mixed model repeated measures; Mean Difference (Net) = 6, 95% CI 2-sided [-82 to 95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 20; Test type: Superiority or Other; p = 0.486, mixed model repeated measures; Mean Difference (Net) = 32, 95% CI 2-sided [-59 to 123] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs Losmapimod 2.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 24; Test type: Superiority or Other; p = 0.604, mixed model repeated measures; Mean Difference (Net) = -24, 95% CI [-113 to 66] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs Losmapimod 7.5 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 24; Test type: Superiority or Other; p = 0.872, mixed model repeated measures; Mean Difference (Net) = -7, 95% CI 2-sided [-97 to 82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs Losmapimod 15 mg; Pre-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 24; Test type: Superiority or Other; p = 0.355, mixed model repeated measures; Mean Difference (Net) = 43, 95% CI 2-sided [-48 to 134] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 4; Test type: Superiority or Other; p = 0.839, mixed model repeated measures; Mean Difference (Net) = 8, 95% CI 2-sided [-65 to 80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 4; Test type: Superiority or Other; p = 0.741, mixed model repeated measures; Mean Difference (Net) = 12, 95% CI 2-sided [-60 to 84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 4; Test type: Superiority or Other; p = 0.056, mixed model repeated measures; Mean Difference (Net) = 71, 95% CI 2-sided [-1.8 to 143] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 8; Test type: Superiority or Other; p = 0.554, mixed model repeated measures; Mean Difference (Net) = -25, 95% CI 2-sided [-107 to 57] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 8; Test type: Superiority or Other; p = 0.472, mixed model repeated measures; Mean Difference (Net) = -30, 95% CI 2-sided [-110 to 51] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 8; Test type: Superiority or Other; p = 0.116, mixed model repeated measures; Mean Difference (Net) = 66, 95% CI 2-sided [-16 to 149] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 12; Test type: Superiority or Other; p = 0.805, mixed model repeated measures; Mean Difference (Net) = -11, 95% CI 2-sided [-98 to 76] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 12; Test type: Superiority or Other; p = 0.763, mixed model repeated measures; Mean Difference (Net) = 13, 95% CI 2-sided [-73 to 100] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 12; Test type: Superiority or Other; p = 0.096, mixed model repeated measures; Mean Difference (Net) = 75, 95% CI 2-sided [-13 to 163] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 16; Test type: Superiority or Other; p = 0.485, mixed model repeated measures; Mean Difference (Net) = -31, 95% CI 2-sided [-118 to 56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 29: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 16; Test type: Superiority or Other; p = 0.704, mixed model repeated measures; Mean Difference (Net) = 17, 95% CI 2-sided [-69 to 103] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 30: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 16; Test type: Superiority or Other; p = 0.108, mixed model repeated measures; Mean Difference (Net) = 72, 95% CI 2-sided [-16 to 159] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 31: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 20; Test type: Superiority or Other; p = 0.147, mixed model repeated measures; Mean Difference (Net) = -64, 95% CI [-151 to 23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 32: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 20; Test type: Superiority or Other; p = 0.792, mixed model repeated measures; Mean Difference (Net) = -12, 95% CI 2-sided [-98 to 75] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 33: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 20; Test type: Superiority or Other; p = 0.275, mixed model repeated measures; Mean Difference (Final Values) = 49, 95% CI [-39 to 138] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 34: Comparison: Placebo vs Losmapimod 2.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 2.5 mg at Week 24; Test type: Superiority or Other; p = 0.530, mixed model repeated measures; Mean Difference (Net) = -28, 95% CI 2-sided [-115 to 59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 35: Comparison: Placebo vs Losmapimod 7.5 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 7.5 mg at Week 24; Test type: Superiority or Other; p = 0.827, mixed model repeated measures; Mean Difference (Net) = 10, 95% CI 2-sided [-77 to 96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 36: Comparison: Placebo vs Losmapimod 15 mg; Post-Bronchodilator FVC for Placebo versus Losmapimod 15 mg at Week 24; Test type: Superiority or Other; p = 0.434, mixed model repeated measures; Mean Difference (Net) = 35, 95% CI 2-sided [-53 to 124] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in St Georges Respiratory Questionnaire for COPD (SGRQ-C) at Week 12 and 24
Description: The SGRQ-C questionnaire had 14 questions of COPD and participant had to rate each question. These 14 questions were separated to evaluate the three components of SGRQ-C. These three components were symptom component (question 1 to 7), activity component (question 9 and 12) and impact component (question 8, 10, 11, 13 and 14). The total score is 0 to 100 with a higher score indicating greater impairment of health status. Change from Baseline was calculated as the specified time point value minus the Baseline value. Baseline visit was Visit 2 (Week 0).
Time Frame: Baseline (Week 0) and Week 12, 24
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
Number analyzed (Participants) | 153 | 149 | 151 | 149
Score on scale
  Week 12: number analyzed (Participants) | 140 | 136 | 139 | 131
  Week 12 | 51.1 (0.98) | 50.6 (0.99) | 52.6 (0.98) | 49.3 (1.01)
  Week 24: number analyzed (Participants) | 131 | 129 | 133 | 121
  Week 24 | 50.6 (1.11) | 51.0 (1.12) | 52.5 (1.10) | 49.2 (1.15)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 12; Test type: Superiority or Other; p = 0.686, mixed model repeated measures; Mean Difference (Net) = -0.6, 95% CI 2-sided [-3.3 to 2.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 12; Test type: Superiority or Other; p = 0.279, mixed model repeated measures; Mean Difference (Net) = 1.5, 95% CI 2-sided [-1.2 to 4.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 12; Test type: Superiority or Other; p = 0.193, mixed model repeated measures; Mean Difference (Net) = -1.8, 95% CI 2-sided [-4.6 to 0.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 24; Test type: Superiority or Other; p = 0.803, mixed model repeated measures; Mean Difference (Net) = 0.4, 95% CI 2-sided [-2.7 to 3.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 24; Test type: Superiority or Other; p = 0.229, mixed model repeated measures; Mean Difference (Net) = 1.9, 95% CI 2-sided [-1.2 to 5.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 24; Test type: Superiority or Other; p = 0.390, mixed model repeated measures; Mean Difference (Net) = -1.4, 95% CI 2-sided [-4.5 to 1.8] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Inspiratory Capacity (IC), Residual Volume(RV), Total Lung Capacity(TLC) , Thoracic Gas Volume (TGV) at Functional Residual Capacity ( FRC), Slow Vital Capacity (SVC) at Week 12 and 24
Description: A plethysmograph is an instrument for measuring changes in volume within an organ or whole body (usually resulting from fluctuations in the amount of blood or air it contains). Plethysmography was used to assess IC, RV, TGV at FRC, SLV, and TLC. Change from Baseline was calculated as the endpoint value minus the Baseline value. Baseline visit was Visit 2 (Week 0).
Time Frame: Baseline(Week 0) and Week 12, 24
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
Number analyzed (Participants) | 153 | 149 | 151 | 149
mL
  IC,Week 12: number analyzed (Participants) | 126 | 130 | 131 | 121
  IC,Week 12 | -26 (34.7) | -4 (34.2) | -80 (34.0) | 13 (35.4)
  IC,Week 24: number analyzed (Participants) | 120 | 126 | 122 | 112
  IC,Week 24 | -9 (39.2) | -53 (38.4) | -62 (38.7) | -50 (40.4)
  RV, Week 12: number analyzed (Participants) | 126 | 130 | 131 | 121
  RV, Week 12 | -14 (69.6) | 21 (68.4) | 13 (68.1) | -43 (70.8)
  RV,Week 24: number analyzed (Participants) | 120 | 126 | 122 | 112
  RV,Week 24 | -127 (74.0) | 11 (72.6) | 72 (73.0) | 5 (76.1)
  TLC, Week 12: number analyzed (Participants) | 126 | 130 | 131 | 121
  TLC, Week 12 | 8 (69.9) | 61 (68.8) | 25 (68.5) | -38 (71.2)
  TLC,Week 24: number analyzed (Participants) | 120 | 126 | 122 | 112
  TLC,Week 24 | -112 (70.2) | -37 (69.0) | 38 (69.3) | -18 (72.3)
  FRC, Week 12: number analyzed (Participants) | 126 | 130 | 131 | 121
  FRC, Week 12 | 24 (68.5) | 61 (67.5) | 92 (67.1) | -43 (69.8)
  FRC, Week 24: number analyzed (Participants) | 120 | 125 | 123 | 112
  FRC, Week 24 | -109 (67.1) | 64 (65.8) | 86 (66.0) | 30 (68.9)
  SVC, Week 12: number analyzed (Participants) | 126 | 130 | 131 | 121
  SVC, Week 12 | 50 (45.8) | 8 (45.0) | -18 (44.8) | 25 (46.5)
  SVC,Week 24: number analyzed (Participants) | 120 | 126 | 122 | 112
  SVC,Week 24 | 27 (52.3) | -93 (51.1) | -10 (51.7) | -7 (53.8)

6. Secondary Outcome: Least Square Mean Ratio to Baseline of Plasma Fibrinogen Over 24 Weeks
Description: Least square mean ratio to Baseline of plasma fibrinogen was assessed at Week 4, 8, 12, 24. Blood samples for biomarker analysis were taken at selected visits.
Time Frame: Baseline (Week 0) and Week 4, 8, 12, 24
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
Number analyzed (Participants) | 153 | 149 | 151 | 149
Ratio
  Week 4: number analyzed (Participants) | 129 | 126 | 138 | 119
  Week 4 | 0.97 (0.022) | 0.96 (0.022) | 0.89 (0.021) | 0.87 (0.022)
  Week 8: number analyzed (Participants) | 123 | 120 | 132 | 115
  Week 8 | 1.01 (0.021) | 0.95 (0.021) | 0.91 (0.020) | 0.89 (0.021)
  Week 12: number analyzed (Participants) | 121 | 112 | 124 | 114
  Week 12 | 0.97 (0.022) | 0.96 (0.022) | 0.89 (0.021) | 0.87 (0.022)
  Week 24: number analyzed (Participants) | 119 | 115 | 124 | 112
  Week 24 | 0.94 (0.021) | 0.94 (0.022) | 0.90 (0.021) | 0.89 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 4; Test type: Superiority or Other; p = 0.157, mixed model repeated measures; Mean Difference (Net) = 0.96, 95% CI 2-sided [0.91 to 1.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 4; Test type: Superiority or Other; p = 0.000, mixed model repeated measures; Mean Difference (Net) = 0.91, 95% CI 2-sided [0.86 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 4; Test type: Superiority or Other; p = 0.000, mixed model repeated measures; Mean Difference (Net) = 0.91, 95% CI 2-sided [0.86 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 8; Test type: Superiority or Other; p = 0.072, mixed model repeated measures; Mean Difference (Net) = 0.95, 95% CI [0.90 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 8; Test type: Superiority or Other; p = 0.000, mixed model repeated measures; Mean Difference (Net) = 0.90, 95% CI 2-sided [0.85 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 8; Test type: Superiority or Other; p = 0.000, mixed model repeated measures; Mean Difference (Net) = 0.88, 95% CI 2-sided [0.83 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 12; Test type: Superiority or Other; p = 0.728, mixed model repeated measures; Mean Difference (Net) = 0.99, 95% CI 2-sided [0.93 to 1.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 12; Test type: Superiority or Other; p = 0.002, mixed model repeated measures; Mean Difference (Net) = 0.91, 95% CI 2-sided [0.86 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 12; Test type: Superiority or Other; p = 0.001, mixed model repeated measures; Mean Difference (Net) = 0.90, 95% CI 2-sided [0.84 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 24; Test type: Superiority or Other; p = 0.823, mixed model repeated measures; Mean Difference (Net) = 1.01, 95% CI 2-sided [0.95 to 1.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 24; Test type: Superiority or Other; p = 0.153, mixed model repeated measures; Mean Difference (Net) = 0.96, 95% CI 2-sided [0.90 to 1.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 24; Test type: Superiority or Other; p = 0.126, mixed model repeated measures; Mean Difference (Net) = 0.95, 95% CI 2-sided [0.90 to 1.01] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Least Square Mean Ratio to Baseline of High Sensitivity C-reactive Protein (HsCRP) Over 24 Weeks
Description: Least square mean ratio to Baseline of HsCRP was assessed at Week 4, 8, 12, 24. Blood samples for biomarker analysis were taken at selected visits.
Time Frame: Baseline (Week 0) and Week 4, 8, 12, 24
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
Number analyzed (Participants) | 153 | 149 | 151 | 149
Ratio
  Week 4: number analyzed (Participants) | 139 | 133 | 141 | 128
  Week 4 | 1.06 (0.089) | 0.93 (0.091) | 0.82 (0.089) | 0.77 (0.091)
  Week 8: number analyzed (Participants) | 144 | 139 | 144 | 137
  Week 8 | 1.02 (0.086) | 1.06 (0.088) | 0.78 (0.085) | 0.75 (0.089)
  Week 12: number analyzed (Participants) | 133 | 126 | 132 | 122
  Week 12 | 1.09 (0.088) | 0.99 (0.090) | 0.79 (0.088) | 0.69 (0.091)
  Week 24: number analyzed (Participants) | 134 | 128 | 131 | 120
  Week 24 | 1.00 (0.088) | 0.95 (0.090) | 0.81 (0.089) | 0.86 (0.093)
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 4; Test type: Superiority or Other; p = 0.291, mixed model repeated measures; Mean Difference (Net) = 0.87, 95% CI 2-sided [0.68 to 1.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 4; Test type: Superiority or Other; p = 0.046, mixed model repeated measures; Mean Difference (Net) = 0.78, 95% CI 2-sided [0.61 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 4; Test type: Superiority or Other; p = 0.014, mixed model repeated measures; Mean Difference (Net) = 0.73, 95% CI 2-sided [0.57 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 8; Test type: Superiority or Other; p = 0.755, mixed model repeated measures; Mean Difference (Net) = 1.04, 95% CI 2-sided [0.82 to 1.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 8; Test type: Superiority or Other; p = 0.029, mixed model repeated measures; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.60 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 7.5 mg at Week 8; Test type: Superiority or Other; p = 0.015, mixed model repeated measures; Mean Difference (Net) = 0.74, 95% CI 2-sided [0.58 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 12; Test type: Superiority or Other; p = 0.468, mixed model repeated measures; Mean Difference (Net) = 0.91, 95% CI 2-sided [0.71 to 1.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 12; Test type: Superiority or Other; p = 0.011, mixed model repeated measures; Mean Difference (Net) = 0.73, 95% CI [0.57 to 0.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 12; Test type: Superiority or Other; p = 0.000, mixed model repeated measures; Mean Difference (Net) = 0.64, 95% CI 2-sided [0.50 to 0.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs Losmapimod 2.5 mg; Placebo versus Losmapimod 2.5 mg at Week 24; Test type: Superiority or Other; p = 0.696, mixed model repeated measures; Mean Difference (Net) = 0.95, 95% CI 2-sided [0.74 to 1.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg at Week 24; Test type: Superiority or Other; p = 0.099, mixed model repeated measures; Mean Difference (Net) = 0.81, 95% CI 2-sided [0.64 to 1.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg at Week 24; Test type: Superiority or Other; p = 0.256, mixed model repeated measures; Mean Difference (Net) = 0.86, 95% CI 2-sided [0.67 to 1.11] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Total Number of Exacerbations Over 24 Weeks
Description: An exacerbation of COPD is defined as a worsening of COPD symptoms requiring changes to normal treatment (other than increased use of relief salbutamol/albuterol) including antimicrobial therapy, short courses of oral steroids, other bronchodilator therapy and/or emergency treatment or hospitalization.
Time Frame: Up to 24 weeks
Population: ITT population.
Measure: Number; unit: Number of exacerbations
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
Number analyzed (Participants) | 153 | 149 | 151 | 149
Number of exacerbations | 48 | 46 | 47 | 34
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 2.5 mg; Losmapimod 2.5 mg versus Placebo; Test type: Superiority or Other; p = 0.989, Negative Binomial regression model; Covariates of treatment, group, smoking status, history of exacerbations and region, with logarithm of time on treatment as an offset variable; Rate ratio = 1.00, 95% CI 2-sided [0.64 to 1.54] — Rate ratio= (Rate of exacerbation in Losmapimod 2.5 mg arm) / (Rate of exacerbation in placebo arm)
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg; Placebo versus Losmapimod 7.5 mg; Test type: Superiority or Other; p = 0.915, Negative Binomial regression model; [statistical method as in outcome 8, analysis 1]; Rate ratio = 0.98, 95% CI [0.64 to 1.50] — Rate ratio= (Rate of exacerbation in Losmapimod 7.5 mg arm) / (Rate of exacerbation in placebo arm)
Statistical Analysis 3: Comparison: Placebo vs Losmapimod 15 mg; Placebo versus Losmapimod 15 mg; Test type: Superiority or Other; p = 0.210, Negative Binomial regression model; [statistical method as in outcome 8, analysis 1]; Rate ratio = 0.74, 95% CI 2-sided [0.47 to 1.18] — Rate ratio= (Rate of exacerbation in Losmapimod 15 mg arm) / (Rate of exacerbation in placebo arm)

ADVERSE EVENTS:
Time Frame: Data for adverse event (AE) was collected up to 1 week after the end of treatment (Week 24) or an early withdrawal visit.
Description: Safety population was used for the analysis of AEs.
Arm/Group | Placebo | Losmapimod 2.5 mg | Losmapimod 7.5 mg | Losmapimod 15 mg
All-Cause Mortality (participants affected / at risk) | 3/153 | 0/149 | 1/151 | 2/149
Serious Adverse Events (participants affected / at risk) | 17/153 | 12/149 | 14/151 | 15/149
Other Adverse Events (participants affected / at risk) | 51/153 | 49/149 | 51/151 | 48/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=153) | Losmapimod 2.5 mg (N=149) | Losmapimod 7.5 mg (N=151) | Losmapimod 15 mg (N=149)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 2 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 1 | 4
Sinobronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Polyp (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=153) | Losmapimod 2.5 mg (N=149) | Losmapimod 7.5 mg (N=151) | Losmapimod 15 mg (N=149)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 30 (35) | 30 (41) | 36 (43) | 24 (32)
Headache (Nervous system disorders) | 13 (24) | 15 (21) | 11 (13) | 13 (19)
Nasopharyngitis (Infections and infestations) | 12 (12) | 8 (9) | 5 (6) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 7 (7) | 5 (6) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.